CLINICAL TRIAL: NCT05155644
Title: Safety of Therapeutic Step-down in Neuromyelitis Optica
Acronym: NMO
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7808
Record Dates: First submitted 2021-10-07; First posted 2021-12-13 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-10

CONDITIONS: Neuromyelitis Optica
Keywords: Neuromyelitis Optica; NMO; multiple sclerosis (MS); Iatrogeny.; Autoimmune diseases
MeSH Terms: conditions — Neuromyelitis Optica; Multiple Sclerosis; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuromyelitis Optica (NMO) is a neuroinflammatory disease related to multiple sclerosis (MS). It affects young subjects and causes a lot of handicap without treatment. Thus, aggressive treatments are frequently introduced early in the life of patients and maintained over the long term. A long duration of treatment exposes to iatrogenism. Therapeutic de-escalation trials in MS or other autoimmune diseases show rebound phenomena. In the NMO, there are no published data on the tolerance of desescalations to guide such strategies.

ELIGIBILITY:
Inclusion criteria:

* Major patients who have received long-term treatment for NMO
* Patients with a prospectively diagnosed NMO using the 2015 NMO classification criteria (IPND)
* Patients who retrospectively meet the classification criteria of the 2015 NMO (IPND)
* Patients who have not expressed their opposition, after information, to the reuse of their data for research purposes.

Exclusion criteria:

* Patient who expressed his opposition to participating in the study
* Lack of data on the assay of anti-AQP4 and anti-MOG antibodies
* Less than a year of taking a second-line treatment before the relay
* End of follow-up <1 year following the transfer, this therefore includes patients whose transfer took place less than one year before the date of data extraction

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major patients who have received long-term treatment for NMO and with a prospectively diagnosed NMO using the 2015 NMO classification criteria (IPND)
Sampling Method: Non-Probability Sample
Enrollment: 947 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Retrospective evaluation of the risk of rebound during therapeutic escalations in neuromyelitis optica (NMO) | Files analysed retrospectively from January 01, 2000 to December 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme DE SÈZE, MD, PhD, Principal Investigator — Service de Neurologie - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Neurologie - Hôpitaux Universitaires de Strasbourg, Strasbourg, France